CLINICAL TRIAL: NCT00356759
Title: A Randomized Double-blind Study of 4-weekly Versus 12-weekly Monitoring of Stable Patients on Long-term Anticoagulation With Warfarin
Brief Title: Prolongation of the Interval Between Monitoring of Warfarin in Stable Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Principal Investigator, Sam Schulman, Prof., McMaster University
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PSI-06-21
Record Dates: First submitted 2006-07-24; First posted 2006-07-26 (Estimated); Results first posted 2018-08-22 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Atrial Fibrillation; Heart Valve Diseases; Venous Thrombosis
Keywords: warfarin; prothrombin time; monitoring
MeSH Terms: conditions — Atrial Fibrillation; Heart Valve Diseases; Venous Thrombosis | interventions — Warfarin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 12-weekly INR (Sham Comparator): Dosing warfarin every 12 weeks, sham INRs 2 out of 3 times
  Interventions: Drug: Dosing warfarin every 12 weeks, sham INRs 2 out of 3 times
- Standard management (No Intervention): Dosing warfarin every 4 weeks, all INRs true values

INTERVENTIONS:
Drug: Dosing warfarin every 12 weeks, sham INRs 2 out of 3 times — Warfarin is dosed according to INR to maintain INR 2.0-3.0 or for mechanical mitral valves or mechanical aortic valves with atrial fibrillation INR 2.5-3.5
  Other Names: warfarin, Coumadin
  Arms: 12-weekly INR

SUMMARY:
Patients with mechanical heart valve prosthesis or with irregular beat (atrial fibrillation) have a high risk of blood clot formation. Such clots can result in a stroke. The patients are treated with warfarin - a "blood thinner" - to prevent these complications. The treatment has to be monitored with a blood test called Prothrombin time (PT) every 1-4 weeks. The dose of warfarin has to be changed whenever the PT result is outside of the treatment range. If the result is too low there is an increased risk of blood clots. If, instead, the result is too high there is a risk of bleeding. One third of the patients have very stable PT results and hardly ever have to change the dose.

The investigators hypothesis is that these patients can go less often, e.g. every 12 weeks, for the blood tests.

DETAILED DESCRIPTION:
OBJECTIVE: The PRolongation of the INTerval between prothrombin time tests in stable patients (PRINT) is a single center, randomized, double-blind study to demonstrate that testing the prothrombin time every 12 weeks provides the same level of anticoagulant control as conventional testing every 4 weeks in this subset of stable patients. This study will enroll patients who have been treated with vitamin K antagonists (VKA) for at least 6 months and have not had any change to the maintenance dose for the most recent 6 months.

HYPOTHESIS: Our hypothesis is that by extending the interval between tests to 12 weeks in these stable patients, the same level of anticoagulant control, can be maintained. With the large and constantly increasing number of patients on warfarin, a reduced frequency of testing would yield considerable savings for the health care system and a decreased burden for the patient. A review of our anticoagulant clinic revealed that one third of the patients would be eligible for such a prolongation of the test interval.

STUDY DESIGN: The proposal is a randomized, double-blind, controlled single centre trial performed at Hamilton Health Sciences - General Hospital. Main inclusion criteria are: long-term anticoagulant therapy, managed by our clinic for at least 6 months and with unchanged maintenance dose for at least 6 months. Eligible and consenting patients identified at annual review visits or from the register of patients monitored by the clinic, will be randomized to dosing of warfarin every 4 weeks (control) or every 12 weeks (experimental). All patients will, however, have blood drawn every 4 weeks. Randomization will be performed using a computer-generated randomization sequence. Stratification is done for the two laboratories performing the analysis and for the two therapeutic ranges that patients are to be maintained within, depending on the indication for anticoagulation. Patients with mechanical mitral valve prosthesis are maintained between 2.5 and 3.5, others between 2.0 and 3.0.The randomization sequence will guide the Coordinating and Methods Center to the correct reporting procedure for each patient, and to provide sham INR-values for two out of each set of three 4-weekly tests in the patients allocated to 12-weekly monitoring. Extreme INR results (<1.5 or >4.4) will always be reported as true results. The investigator and the patient are blind to the procedure and are only aware of the sequence order number.The patients are carefully instructed about risk factors that can change the effect of VKA. They are contacted by telephone after each test for information on the result, the dosing and for questioning of adverse events. After 12 months in the study there is a final visit scheduled at the anticoagulation clinic for review of the patient.

ANALYSIS: After the last patient has concluded the study, all clinical data will be transferred to the study statistician for analysis. The primary outcome measure is "the time in therapeutic range" (TTR). The secondary outcome measures are "proportion of patients with extreme INR results", "proportion of INR results that are extreme" and "number of changes of the maintenance dose". These are well-recognized tools for evaluation of the level of anticoagulant control. Major bleeding and objectively verified thromboembolic events will also be registered, but the expected number is very small and not sufficient for any statistical analyses.

SAMPLE SIZE: Sample size calculations are based on 77% TTR for a population with very stable VKA-dose and a maximum tolerable deviation of 7.5 percentage points; one-sided alpha of 2.5% and power of 90%. The sample will accordingly be 107 patients per group. After interim analysis the DSMB recommended to expand the sample size to 125 patients per group (July 16, 2008).

ELIGIBILITY:
Inclusion Criteria:

* Patients on long-term warfarin (for prophylaxis of arterial embolism in patients with atrial fibrillation or mechanical heart valve replacement, or secondary prophylaxis after VTE) with a target INR of 2.0-3.0 or 2.5-3.5,
* Anticoagulant therapy managed by the clinic (HHS - General Hospital) for at least 6 months prior to enrolment, and
* Maintenance dose of warfarin unchanged for the previous 6 months or longer.

Exclusion Criteria:

* Age <18 years,
* Life expectancy of less than 1 year,
* Attending physician believes the patient is not suitable for the study (e.g. psychiatric disorder, history of non-compliance),
* Geographic inaccessibility or
* Failure to obtain written consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2006-12; Primary Completion 2010-01 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sam Schulman, Professor, Principal Investigator — McMaster University
Locations (1):
- HHS - General Hospital, Thrombosis Service, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schulman S, Parpia S, Stewart C, Rudd-Scott L, Julian JA, Levine M. Warfarin dose assessment every 4 weeks versus every 12 weeks in patients with stable international normalized ratios: a randomized trial. Ann Intern Med. 2011 Nov 15;155(10):653-9, W201-3. doi: 10.7326/0003-4819-155-10-201111150-00003. PMID 22084331

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Assessment 4-weekly: INRs and dose assessments every 4 weeks true values, no sham INRs
- Dose Assessment 12-weekly: INRs and dose assessment 4-weekly, but 2 of 3 INRs are sham results, so dose assessment on true result is only 12-weekly
Period: Overall Study
Arm/Group | Dose Assessment 4-weekly | Dose Assessment 12-weekly
Started | 126 | 124
Completed | 112 | 114
Not Completed | 14 | 10
Not completed — Death | 5 | 2
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Adverse Event | 1 | 3
Not completed — Lost to Follow-up | 1 | 1
Not completed — Intercurrent disease or persistent extre | 5 | 2

BASELINE CHARACTERISTICS:
Population: All patients randomized
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Assessment 4-weekly | Dose Assessment 12-weekly | Total
Number analyzed (Participants) | 126 | 124 | 250
Age, Continuous [Median (Full Range); unit: years]
  Age | 72 [29 to 93] | 70 [23 to 92] | 71 [23 to 93]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 37 | 76
  Male | 87 | 87 | 174
Therapeutic INR range [Number; unit: participants] — International normalized ratio (INR) is a standardized expression of the prothrombin time. Normal is 0.9-1.2. Therapeutic range is 2.0-3-0 for most patients, 2.5-3.5 for those with mechanical mitral valve or with mechanical aortic valve plus atrial fibrillation
  participants
    INR range 2.0-3.0 | 111 | 109 | 220
    INR range 2.5-3.5 | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Primary Outcome Measure: Time in Therapeutic Range
Description: Percent time in therapeutic range calculated by linear interpolation.
Time Frame: 12 months
Population: Intention to treat population
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Dose Assessment 4-weekly | Dose Assessment 12-weekly
Number analyzed (Participants) | 126 | 124
percentage of time | 74.1 (18.8) | 71.6 (20.0)

2. Secondary Outcome: Secondary Efficacy Outcomes: Thromboembolic Events
Description: Number of patients with any objectively verified, independently adjudicated thromboembolic event during the 12-month study period
Time Frame: 12 months
Population: Intention to treat
Measure: Number; unit: participants
Arm/Group | Dose Assessment 4-weekly | Dose Assessment 12-weekly
Number analyzed (Participants) | 126 | 124
participants | 1 | 0

3. Secondary Outcome: Secondary Safety Outcome: Major Bleeding
Description: Number of patients with any objectively verified, independently adjudicated major bleeding event during the 12-month study period. Major bleeding was defined according to the International Society on Thrombosis and Haemostasis (ISTH) criteria
Time Frame: 12 months
Population: Intention to treat
Measure: Number; unit: participants
Arm/Group | Dose Assessment 4-weekly | Dose Assessment 12-weekly
Number analyzed (Participants) | 126 | 124
participants | 1 | 2

4. Secondary Outcome: Secondary Safety Outcome: Number of Patients With Extreme INR Results
Description: Secondary safety outcome is number of patients with at least one INR below 1.5 or above 4.4
Time Frame: 12 months
Population: Intention to treat
Measure: Number; unit: participants
Arm/Group | Dose Assessment 4-weekly | Dose Assessment 12-weekly
Number analyzed (Participants) | 126 | 124
participants | 27 | 19

5. Secondary Outcome: Number of Extreme INR Results
Description: Number of INRs outside the range 1.5-4.4
Time Frame: 12 months
Population: Intention to treat
Measure: Number; unit: Number of tests
Arm/Group | Dose Assessment 4-weekly | Dose Assessment 12-weekly
Number analyzed (Participants) | 126 | 124
Number of tests | 27 | 17

6. Secondary Outcome: Patients With Dose Changes
Description: Number of patients with at least one change of maintenance dose during the 12-month study period
Time Frame: 12 months
Population: Intention to treat
Measure: Number; unit: participants
Arm/Group | Dose Assessment 4-weekly | Dose Assessment 12-weekly
Number analyzed (Participants) | 126 | 124
participants | 70 | 46

ADVERSE EVENTS:
Time Frame: 12 months
Description: Fatal events are reported as serious adverse events. Non-fatal major bleeding or thromboembolism are reported as serious adverse events. Minor bleeding events are reported as non-serious (other) adverse events.
Groups:
- 12-weekly INR: Patients had INR every 4 weeks but only every thisrd INR was true; the other two were sham INRs dampened to be within or close to therapeutic range. Thus, true dose assessment was in practice performed every 12 weeks
- 4-weekly INR: Patients had INR every 4 weeks and all results were true. Thus, true dose assessments were performed every 4 weeks.
Arm/Group | 12-weekly INR | 4-weekly INR
All-Cause Mortality (participants affected / at risk) | 2/124 | 5/126
Serious Adverse Events (participants affected / at risk) | 4/124 | 7/126
Other Adverse Events (participants affected / at risk) | 7/124 | 4/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 12-weekly INR (N=124) | 4-weekly INR (N=126)
Cardiac death (Cardiac disorders) | 1 (1) | 3 (3)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) — Pancreatitis with fatal septic shock
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) — Fatal respiratory failure
Gastrointestinal bleeding (Gastrointestinal disorders) | 2 (2) | 1 (1) — Melena
Renal infarct (Renal and urinary disorders) | 0 (0) | 1 (1) — Arterial embolism
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 12-weekly INR (N=124) | 4-weekly INR (N=126)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) — Bleeding from the nose that did not fulfill criteria for major bleeding
Hematuria (Renal and urinary disorders) | 2 (2) | 1 (1) — Urinary tract bleeding that did not meet criteria for major bleeding
Rectal bleeding (Gastrointestinal disorders) | 1 (1) | 1 (1) — Bleeding from rectum bleeding that did not meet criteria for major bleeding
Subconjunctival bleeding (Eye disorders) | 0 (0) | 1 (1) — Subconjunctival eye bleeding that did not meet criteria for major bleeding

LIMITATIONS AND CAVEATS:
Not a truly INR monitoring and dosing every 12 weeks, because patients were tested and contacted every 4 weeks for sham results and to remind of important factors for INR instability. Extreme INR results in the 12-week group were reported unblinded.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes